CLINICAL TRIAL: NCT05190952
Title: A Comparative Study Between Dexamethasone and Ketamine as Adjuvants to Bupivacaine for Incisional Infiltration in Pediatric Abdominal Operations
Brief Title: Dexamethasone & Ketamine as Adjuvants to Bupivacaine for Incisional Infiltration in Pediatric Abdominal Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Diaaeldein Mahmoud Haiba, Lecturer of Anesthesia, ICU & Pain management, Faculty of medicine, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R 122A/2020
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Pediatric ALL
Keywords: bupivacine; Ketamine; dexamethasone
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Bupivacaine; Ketamine; Dexamethasone

STUDY DESIGN:
Intervention Model Description: a randomized, controlled, double blind study
Who Masked: Participant, Investigator
Masking Description: Both the patient and the attending anesthesiologist will be blinded to the drugs injected (a randomized, controlled, double blind study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Control Group (Bupivacaine 0.25% 1ml/kg will be injected subcutaneously by the surgeon before wound closure).
  Interventions: Drug: Bupivacaine
- Group 2 (Active Comparator): Ketamine Group (In addition to bupivacaine, ketamine 1mg/kg diluted in 10 ml normal saline will be injected subcutaneously by the surgeon before wound closure. Bupivacaine and ketamine will be administered using two separate syringes).
  Interventions: Drug: Bupivacaine; Drug: Ketamine
- Group 3 (Active Comparator): Dexamethasone Group (In addition to bupivacaine, dexamethasone 0.2mg/kg diluted in 10 ml normal saline will be injected subcutaneously by the surgeon before wound closure. Bupivacaine and dexamethsone will be administered using two separate syringes).
  Interventions: Drug: Bupivacaine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine 0.25% 1ml/kg will be injected subcutaneously by the surgeon before wound closure.
Drug: Ketamine — In addition to bupivacaine, ketamine 1mg/kg diluted in 10 ml normal saline will be injected subcutaneously by the surgeon before wound closure. Bupivacaine and ketamine will be administered using two separate syringes.
  Arms: Group 2
Drug: Dexamethasone — In addition to bupivacaine, dexamethasone 0.2mg/kg diluted in 10 ml normal saline will be injected subcutaneously by the surgeon before wound closure. Bupivacaine and dexamethsone will be administered using two separate syringes.
  Arms: Group 3

SUMMARY:
The aim of this study is to compare the effects of both ketamine and dexamethasone on the duration and magnitude of analgesia when combined with bupivacaine for incisional infiltration in pediatric abdominal operations.

DETAILED DESCRIPTION:
Wound infiltration with local anaesthetics is a simple, effective and inexpensive means of providing good analgesia for a variety of surgical procedures without any major side-effects.

Patients and Methods Type of Study:Randomized, controlled, double-blind study.

Study Setting: Ain Shams university hospitals.

Study Period: 3months after approval of the ethical committee.

Study Population:

Inclusion Criteria:

Children of both sexes aged 1-8 years, ASA I-II, undergoing moderate to major abdominal operations.

Exclusion Criteria:

History of diabetes, cardiac or neurological disease Hypersensitivity to any of the drugs used in the study Risk of wound complications ( as infected wound, history of wound dehiscence, hypo-albuminaemia) Multiple incision sites Operations scheduled as day-case

Sample size: using PASS program version 15, setting alpha error at 5%and power at 80%. Based on previous studies the needed sample is 50 cases per group (total 150 patients).

Sampling Method: simple random sampling Children will be randomized into three groups 50 patients each.

* Group I: Bupivacaine 0.25% 1ml/kg will be injected subcutaneously by the surgeon before wound closure.
* Group II: In addition to bupivacaine, ketamine 1mg/kg diluted in 10 ml normal saline will be injected subcutaneously by the surgeon before wound closure. Bupivacaine and ketamine will be administered using two separate syringes.
* Group III: In addition to bupivacaine, dexamethasone 0.2mg/kg diluted in 10 ml normal saline will be injected subcutaneously by the surgeon before wound closure. Bupivacaine and dexamethsone will be administered using two separate syringes.

Study Tools and Study Procedures:

In all groups, drugs will be prepared by the attending anesthesiologist and injected by the surgeon (both will be blinded to the procedure) Anesthetic technique In all children, anesthesia will be induced by sevoflurane or propofol 2mg/kg IV, fentanyl 2ug/kg, atracurium 0.5 mg/kg followed by endotracheal intubation and mechanical ventilation with pressure controlled mode. Anesthesia will be maintained with sevoflurane in oxygen. All children will be monitored using ECG, non invasive blood pressure cuff, pulse oximeter and temperature probe. Ringer acetate will be used as the replacement fluid. At conclusion of surgery, the trachea will be extubated after reversal of the muscle relaxant with neostigmine 0.05 mg/kg + atropine 0.02 mg/kg and the child transferred to the postanesthesia care unit.

Comparisons will be done between both groups as regards: time needed for first analgesic dose (primary outcome), The FLACC pain scale will be assesed over a 24hour period as follows: (table 1) in PACU, then 2 hourly for 12 hours then 4 hourly.),Total number of administrations of rescue analgesia in the first 24 hours postoperatively, incidence of wound complications over a 7 d period (secondary outcomes)

First analgesic dose:

If the FLACC scale was more than 3 either during intervals of FLACC recording or in between, intravenous paracetamol was provided at a dose of 15mg/kg then fixed around the clock every 6 hours.

Rescue analgesia If pain persisted or recurred rectal diclophenac 1mg/kg or ibuprophen in children in whom oral intake has been allowed.

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes aged 1-8 years, ASA I-II, undergoing moderate to major abdominal operations.

Exclusion Criteria:

* History of diabetes, cardiac or neurological disease
* Hypersensitivity to any of the drugs used in the study.
* Risk of wound complications ( as infected wound, history of wound dehiscence, hypo--albuminaemia)
* Multiple incision sites

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2020-12-05 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
The Face, Leg, Activity, Cry and Consolability scale (FLACC) pain scale | At Time zero (The time of extubation)
  -Face: No particular expression or smile (0) Occasional grimace or frown, withdrawn, disinterested (1) Frequent to constant frown, clenched jaw, quivering chin (2)
  -Legs: Normal position or relaxed (0) Uneasy, restless, tense (1) Kicking, legs drawn up (2)
  -Activity: Lying quietly, normal position, moves easily (0) Squirming, shifting back and forth, tense (1) Arched, rigid or jerking (2)
  -Cry: No crying (awake or asleep) (0) Moans or whimpers, occasional complaint (1) Crying steadily, screamsor sobs, frequent complaints (2)
  -Consolability: Content, relaxed (0) Reassured by occasional touching, hugging or talking to, distractable (1) Difficult to console or comfort (2)
  The scale range from 0 to 10. The higher the number the worse the pain status.
The Face, Leg, Activity, Cry and Consolability scale (FLACC) pain scale | At 2 hours postoperatively
  -Face: No particular expression or smile (0) Occasional grimace or frown, withdrawn, disinterested (1) Frequent to constant frown, clenched jaw, quivering chin (2)
  -Legs: Normal position or relaxed (0) Uneasy, restless, tense (1) Kicking, legs drawn up (2)
  -Activity: Lying quietly, normal position, moves easily (0) Squirming, shifting back and forth, tense (1) Arched, rigid or jerking (2)
  -Cry: No crying (awake or asleep) (0) Moans or whimpers, occasional complaint (1) Crying steadily, screamsor sobs, frequent complaints (2)
  -Consolability: Content, relaxed (0) Reassured by occasional touching, hugging or talking to, distractable (1) Difficult to console or comfort (2)
  The scale range from 0 to 10. The higher the number the worse the pain status.
The Face, Leg, Activity, Cry and Consolability scale (FLACC) pain scale | At 12 hours postoperatively
  Face:
  No particular expression or smile (0) Occasional grimace or frown, withdrawn, disinterested (1) Frequent to constant frown, clenched jaw, quivering chin (2) -Legs: Normal position or relaxed (0) Uneasy, restless, tense (1) Kicking, legs drawn up (2)
  -Activity: Lying quietly, normal position, moves easily (0) Squirming, shifting back and forth, tense (1) Arched, rigid or jerking (2)
  -Cry: No crying (awake or asleep) (0) Moans or whimpers, occasional complaint (1) Crying steadily, screamsor sobs, frequent complaints (2)
  -Consolability: Content, relaxed (0) Reassured by occasional touching, hugging or talking to, distractable (1) Difficult to console or comfort (2)
  The scale range from 0 to 10. The higher the number the worse the pain status.
The Face, Leg, Activity, Cry and Consolability scale (FLACC) pain scale | At 24 hours postoperatively
  Face:
  No particular expression or smile (0) Occasional grimace or frown, withdrawn, disinterested (1) Frequent to constant frown, clenched jaw, quivering chin (2) -Legs: Normal position or relaxed (0) Uneasy, restless, tense (1) Kicking, legs drawn up (2)
  -Activity: Lying quietly, normal position, moves easily (0) Squirming, shifting back and forth, tense (1) Arched, rigid or jerking (2)
  -Cry: No crying (awake or asleep) (0) Moans or whimpers, occasional complaint (1) Crying steadily, screamsor sobs, frequent complaints (2)
  -Consolability: Content, relaxed (0) Reassured by occasional touching, hugging or talking to, distractable (1) Difficult to console or comfort (2)
  The scale range from 0 to 10. The higher the number the worse the pain status.
Rescue analgesia | 24 hours
  Time needed for first rescue analgesia
Total dose of rescue analgesia in the first 24 hours postoperatively. | 24 hours
  Total dose of rescue analgesia in the first 24 hours postoperatively. If pain persisted or recurred rectal diclophenac 1mg/kg. total dose measured in milligrams

SECONDARY OUTCOMES:
Incidence of wound complications | 72 hours
  Incidence of wound infection or dehiscence, descirbed in the form of occured or not occured.
Incidence of postoperative nausea and vomiting | 24 hours
  Incidence of postoperative nausea and vomiting discribed in the form of occured or not occured

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university hospitals, Cairo, Al Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided